CLINICAL TRIAL: NCT04575753
Title: Evaluating the Role of Pre-existing Resolvins in the Resolution of ICU Delirium
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: CHU de Charleroi (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Anesthesiologist, principal investigator, Université Libre de Bruxelles
Other Study IDs: Resolvin-delirium
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Study group — Blood samples will be taken from ICU patients on the day of ICU admission, day 2 and day 5 after ICU admission.
  Similarly, patients will be subjected to cognitive testing (CAM-ICU) to determine the presence of delirium

SUMMARY:
As patient management is improving, more and more ICU survivors are being confronted with cognitive dysfunction and this well after their hospital stay.

In the ICU, delirium rates have been reported to be as high at 81%. Delirium is associated with patient and family stress, increased hospital costs, increased duration of stay, escalation of care and increased mortality and morbidity.

The physiopathology of ICU cognitive impairment is complex and involves an inflammatory cascade Recently, the role of 'resolvins' derived from omega-3 fatty acids has been studied in the resolution of inflammation.

Therefore, this hypothesis of this study is that ICU patients with higher serum levels of resolvins at ICU admission, ICU day 2 and day 5 will have a lesser degree of cognitive impairment on day 5 of ICU stay.

DETAILED DESCRIPTION:
As patient management is improving, more and more ICU survivors are being confronted with cognitive dysfunction and this well after their hospital stay.

Delirium is characterized by an acute onset or fluctuating course, inattention and either disorganized thought (manifesting as memory, language and orientation difficulties) or altered level of consciousness. Multiple forms exist: hyperactive versus hypoactive versus mixed.

In the ICU, delirium rates have been reported to be as high at 81%. Delirium is associated with patient and family stress, increased hospital costs, increased duration of stay, escalation of care and increased mortality and morbidity.

The physiopathology of ICU cognitive impairment is complex. One theory is that, during infection/trauma, the alarmin high molecular group box 1 (HMGB1) is released into the bloodstream by activated platelets.

This damage-associated molecular pattern (DAMP) can bind to pattern recognition receptors on circulating bone marrow-derived monocytes (BM-DMs), causing a platelet-monocyte interaction but also triggering the nuclear translocation of the transcription factor NF-kappaB which activates gene expression and release of pro-inflammatory cytokines. The onset of this inflammatory state disrupts the blood brain barrier.

Within the brain parenchyma the chemokine MCP-1 and, by signaling through its receptor, CCR2, attracts the BM-DMs. The influx of BM-DMs activates the resident quiescent microglia. Together, BM-DMs and activated microglia release HMGB1, IL-6, and IL-1β ; thereby disrupting long-term potentiation and the synaptic plasticity involved in cognitive functions of learning and memory.

Inability to successfully resolve the inflammatory cascade promotes the development of cognitive impairment.

Recently, the role of 'resolvins' derived from omega-3 fatty acids has been studied in the resolution of inflammation.

In a mouse model of perioperative neurocognitive disorder, maresin 1 (a metabolite of omega-3) improved post-operative cognition and prevented surgery-induced glial activation and opening of the blood brain barrier. Similarly, in the same model, aspirine-triggered resolving D1 improved post-operative cognition, reduced systemic IL-6 levels and reserved surgery-induced astrogliosis.

Mechanically ventilated ICU patients who benefitted from omega-3 supplements, had a lesser degree of ICU delirium.

Therefore, the hypothesis of this study is that ICU patients with higher serum levels of resolvins at ICU admission, ICU day 2 and day 5 will have a lesser degree of cognitive impairment on day 5 of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Non-ventilated, non-sedated adult patients with a planned ICU stay >72 hours. - - patients admitted due to an exacerbation of COPD
* patients admitted due to severe trauma
* patients admitted due to cardiogenic shock
* patients admitted due to septic shock

Exclusion Criteria:

* Patients who don't understand English, French or Dutch
* Patients who are visually/auditory impaired (without glasses/ hearing aid)
* Patients with known neuro-psychiatric disorders
* Patients with known recreational drug and alcohol (ab)use
* Patients with a neurological trauma
* Patients on ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-ventilated, non-sedated adult patients of all genders with a planned ICU stay >72 hours at the CHU de Charleroi, Charleroi, Belgium between October 2020- May 2021 will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The influence of serum levels of resolvins (RvD1) at ICU admission, and ICU day 2 and day 5 on cognitive impairment (defined by CAM-ICU) on day 5 of ICU stay. | 5 days
  Blood samples will be drawn at the day of ICU admission, day 2 and day 5 after ICU admission to measure resolvins (RvD1; 17SHDHA; DHA) through mass spectrometry.
  At the same timepoints, cognitive testing will be performed (CAM-ICU) to determine the presence or absence of delirium on day 5 of ICU admission.
The influence of serum levels of resolvins (DHA) at ICU admission, and ICU day 2 and day 5 on cognitive impairment (defined by CAM-ICU) on day 5 of ICU stay. | 5 days
  Blood samples will be drawn at the day of ICU admission, day 2 and day 5 after ICU admission to measure resolvins (RvD1; 17SHDHA; DHA) through mass spectrometry.
  At the same timepoints, cognitive testing will be performed (CAM-ICU) to determine the presence or absence of delirium on day 5 of ICU admission.
The influence of serum levels of resolvins (17SHDHA)) at ICU admission, and ICU day 2 and day 5 on cognitive impairment (defined by CAM-ICU) on day 5 of ICU stay. | 5 days
  Blood samples will be drawn at the day of ICU admission, day 2 and day 5 after ICU admission to measure resolvins (RvD1; 17SHDHA; DHA) through mass spectrometry.
  At the same timepoints, cognitive testing will be performed (CAM-ICU) to determine the presence or absence of delirium on day 5 of ICU admission.

SECONDARY OUTCOMES:
Inflammatory markers-delirium-day0 | 1 day
  The influence of serum levels of CRP (at ICU admission) on cognitive impairment (defined by CAM-ICU) at ICU admission.
Inflammatory markers-delirium-day0 | 1 day
  The influence of serum levels of TNF-alpha (at ICU admission) on cognitive impairment (defined by CAM-ICU) at ICU admission.
Inflammatory markers-delirium-day0 | 1 day
  The influence of serum levels of HMGB1 (at ICU admission) on cognitive impairment (defined by CAM-ICU) at ICU admission.
Inflammatory markers-delirium-day0 | 1 day
  The influence of serum levels of PF4 (at ICU admission) on cognitive impairment (defined by CAM-ICU) at ICU admission.
Inflammatory markers-delirium-day0 | 1 day
  The influence of serum levels of lactate (at ICU admission) on cognitive impairment (defined by CAM-ICU) at ICU admission.
Inflammatory markers-delirium-day2 | 2 days
  The influence of serum levels of CRP (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers-delirium-day2 | 2 days
  The influence of serum levels of TNF-alpha (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers-delirium-day2 | 2 days
  The influence of serum levels of HMGB1 (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers-delirium-day2 | 2 days
  The influence of serum levels of PF4 (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers-delirium-day2 | 2 days
  The influence of serum levels of lactate (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers-delirium-day5 | 5 days
  The influence of serum levels of CRP (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers-delirium-day5 | 5 days
  The influence of serum levels of TNF-alpha (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers-delirium-day5 | 5 days
  The influence of serum levels of HMGB1 (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers-delirium-day5 | 5 days
  The influence of serum levels of PF4 (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers-delirium-day5 | 5 days
  The influence of serum levels of lactate (at ICU admission) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers2-delirium-2 | 2 days
  The influence of serum levels of CRP (on day 2) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers2-delirium-2 | 2 days
  The influence of serum levels of TNF-alpha (on day 2) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers2-delirium-2 | 2 days
  The influence of serum levels of HMGB1 (on day 2) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers2-delirium-2 | 2 days
  The influence of serum levels of lactate (on day 2) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers2-delirium-2 | 2 days
  The influence of serum levels of PF4 (on day 2) on cognitive impairment (defined by CAM-ICU) on ICU day 2.
Inflammatory markers2-delirium-5 | 5 days
  The influence of serum levels of CRP (on day 2) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers5-delirium-5 | 5 days
  The influence of serum levels of TNF-alpha (on day 5) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers5-delirium-5 | 5 days
  The influence of serum levels of HMGB1 (on day 5) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers5-delirium-5 | 5 days
  The influence of serum levels of PF4 (on day 5) on cognitive impairment (defined by CAM-ICU) on ICU day 5.
Inflammatory markers5-delirium-5 | 5 days
  The influence of serum levels of lactate (on day 5) on cognitive impairment (defined by CAM-ICU) on ICU day 5.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Piagnerelli, MD; PHD, Study Chair — CHU de Charleroi, Belgium
Locations (1):
- CHU-Charleroi Hopital Civil Marie Curie, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will be made available, anonymously, if needed

REFERENCES:
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Leslie DL, Inouye SK. The importance of delirium: economic and societal costs. J Am Geriatr Soc. 2011 Nov;59 Suppl 2(Suppl 2):S241-3. doi: 10.1111/j.1532-5415.2011.03671.x. PMID 22091567
- [Background] Rouhiainen A, Imai S, Rauvala H, Parkkinen J. Occurrence of amphoterin (HMG1) as an endogenous protein of human platelets that is exported to the cell surface upon platelet activation. Thromb Haemost. 2000 Dec;84(6):1087-94. PMID 11154118
- [Background] Vacas S, Degos V, Tracey KJ, Maze M. High-mobility group box 1 protein initiates postoperative cognitive decline by engaging bone marrow-derived macrophages. Anesthesiology. 2014 May;120(5):1160-7. doi: 10.1097/ALN.0000000000000045. PMID 24162463
- [Background] Hu J, Feng X, Valdearcos M, Lutrin D, Uchida Y, Koliwad SK, Maze M. Interleukin-6 is both necessary and sufficient to produce perioperative neurocognitive disorder in mice. Br J Anaesth. 2018 Mar;120(3):537-545. doi: 10.1016/j.bja.2017.11.096. Epub 2018 Feb 3. PMID 29452810
- [Background] Terrando N, Eriksson LI, Ryu JK, Yang T, Monaco C, Feldmann M, Jonsson Fagerlund M, Charo IF, Akassoglou K, Maze M. Resolving postoperative neuroinflammation and cognitive decline. Ann Neurol. 2011 Dec;70(6):986-995. doi: 10.1002/ana.22664. PMID 22190370
- [Background] Cibelli M, Fidalgo AR, Terrando N, Ma D, Monaco C, Feldmann M, Takata M, Lever IJ, Nanchahal J, Fanselow MS, Maze M. Role of interleukin-1beta in postoperative cognitive dysfunction. Ann Neurol. 2010 Sep;68(3):360-8. doi: 10.1002/ana.22082. PMID 20818791
- [Background] Feng X, Valdearcos M, Uchida Y, Lutrin D, Maze M, Koliwad SK. Microglia mediate postoperative hippocampal inflammation and cognitive decline in mice. JCI Insight. 2017 Apr 6;2(7):e91229. doi: 10.1172/jci.insight.91229. PMID 28405620
- [Background] Saxena S, Lai IK, Li R, Maze M. Neuroinflammation is a putative target for the prevention and treatment of perioperative neurocognitive disorders. Br Med Bull. 2019 Jun 19;130(1):125-135. doi: 10.1093/bmb/ldz010. PMID 31049563
- [Background] Ishihara T, Yoshida M, Arita M. Omega-3 fatty acid-derived mediators that control inflammation and tissue homeostasis. Int Immunol. 2019 Aug 23;31(9):559-567. doi: 10.1093/intimm/dxz001. PMID 30772915
- [Background] Yang T, Xu G, Newton PT, Chagin AS, Mkrtchian S, Carlstrom M, Zhang XM, Harris RA, Cooter M, Berger M, Maddipati KR, Akassoglou K, Terrando N. Maresin 1 attenuates neuroinflammation in a mouse model of perioperative neurocognitive disorders. Br J Anaesth. 2019 Mar;122(3):350-360. doi: 10.1016/j.bja.2018.10.062. Epub 2018 Dec 28. PMID 30770053
- [Background] Terrando N, Gomez-Galan M, Yang T, Carlstrom M, Gustavsson D, Harding RE, Lindskog M, Eriksson LI. Aspirin-triggered resolvin D1 prevents surgery-induced cognitive decline. FASEB J. 2013 Sep;27(9):3564-71. doi: 10.1096/fj.13-230276. Epub 2013 May 24. PMID 23709617
- [Background] Naghibi T, Shafigh N, Mazloomzadeh S. Role of omega-3 fatty acids in the prevention of delirium in mechanically ventilated patients. J Res Med Sci. 2020 Jan 20;25:10. doi: 10.4103/jrms.JRMS_567_18. eCollection 2020. PMID 32055250